CLINICAL TRIAL: NCT05414409
Title: The Gut Microbiome in Lean and Overweight Youth With Type 1 Diabetes and Novel Mechanism of Action of Metformin
Brief Title: The Gut Microbiome in Type 1 Diabetes and Mechanism of Metformin Action
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heba M. Ismail (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Heba M. Ismail, Assistant Professor of Pediatrics, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15498; 1K23DK129799 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The investigators will examine the differences in the gut microbiome between lean and overweight/obese youth with type 1 diabetes and then enroll the overweight/obese youth with type 1 diabetes into the clinical trial to receive metformin as an intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparison of microbiome by BMI Category (No Intervention): The gut microbiome and metabolites of 42 lean and 42 overweight/obese youth with type 1 diabetes will be evaluated cross-sectionally.
- Metformin (Experimental): This is a group of 30 youth with type 1 diabetes and overweight/obesity who will receive metformin for 6 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is an oral medication that improves insulin sensitivity.
  Arms: Metformin

SUMMARY:
Ovwerweight and obesity prevalence in persons with T1D has increased, which further complicates management and risk for complications. The proposed study is relevant to public health because it helps us understand the role of the gut microbiome in disease pathophysiology in T1D youth with overweight and obesity as well as potential mechanisms to modify disease.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight/obese youth 11-18 years of age with T1D at time of enrollment.
2. Lean youth 11-18 years of age with T1D at time of enrollment.

Exclusion Criteria:

1. Known monogenic forms of diabetes or Type 2 diabetes (confirmed clinically and by genetic/antibody testing).
2. History of ongoing infection or antibiotic treatment within the past month;
3. History of immune-compromise, recurrent infections, steroid intake (inhaled or oral forms) or other immunosuppressant use in the past 6 months.
4. History of chronic gastrointestinal disease and active within the past 6 months, possible or confirmed celiac disease.
5. Participation in any research intervention trials within the past 3 months.
6. History of treatment or use of metformin, a type 2 diabetes medication.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Differences in the gut microbiome in lean and overweight/obese youth with type 1 diabetes | Baseline
  cross sectional comparison of stool microbiome using metagenomic sequencing data
Differences in the gut microbial metabolites in lean and overweight/obese youth with type 1 diabetes | Baseline
  The investigators will measure and compare the stool and serum short chain fatty acids using mass spectrometry
Differences in the gut microbial metabolites in lean and overweight/obese youth with type 1 diabetes | Baseline
  The investigators will measure and compare the stool and serum secondary bile acids using mass spectrometry
Changes in the gut microbiome in overweight/obese youth with type 1 diabetes in response to metformin | Baseline, Month 3, and Month 6
  longitudinal comparison before and after taking metformin for 6 months, stool samples will be collected at baseline, 3 months and 6 months and sequenced for microbiome profile using metagenomic sequencing
Changes in the gut microbial metabolites in overweight/obese youth with type 1 in response to metformin | Baseline, Month 3, and Month 6
  The investigators will measure and compare the stool and serum metabolites (short chain fatty acids and secondary bile acids) before, during and after 6 months of daily metformin therapy using mass spectrometry

SECONDARY OUTCOMES:
Differences in measures of C-peptide as a measure of beta cell health in lean and overweight/obeseT1D youth | Baseline
  The investigators will measure serum C-peptide to calculate a ratio of proinsulin to C-peptide as a marker of beta cell health. These measures will then be compared between the lean and obese T1D youth.
Differences in measures Proinsulin as a measure of beta cell health in lean and overweight/obeseT1D youth | Baseline
  The investigators will measure serum proinsulin and calculate a ratio of proinsulin to C-peptide as a marker of beta cell health. These measures will then be compared between the lean and obese T1D youth.
Differences in measures of insulin sensitivity in lean and overweight/obese T1D youth | Baseline
  Insulin sensitivity will be assessed in individuals using the estimated insulin sensitivity score (eIS), which is based on waist circumference (cm), HbA1c (%) and triglycerides (mg/dl)
Changes in measures of C-peptide as a measure of beta cell health in overweight/obese T1D youth in response to metformin | Baseline, Month 3, and Month 6
  Serum C-peptide will be used to calculate proinsulin to C-peptide ratio as a measure of beta cell health before and after metformin therapy
Changes in measures of proinsulin as a measure of beta cell health in overweight/obese T1D youth in response to metformin | Baseline, Month 3, and Month 6
  Serum proinsulin will be used to calculate proinsulin to C-peptide ratio as a measure of beta cell health before and after metformin therapy
Changes in measures of insulin sensitivity in overweight/obese T1D youth in response to metformin | Baseline, Month 3, and Month 6
  Estimated insulin sensitivity score will be used to assess response metformin therapy
Changes in measures of beta cell function using a timed mixed meal tolerance test | Baseline and Month 6
  Participants in the metformin trial will undergo a standard 2-hour mixed meal tolerance test at baseline and after 6 months of oral metformin therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No